CLINICAL TRIAL: NCT04367116
Title: The Study to Evaluate the Safety and Efficacy of Spinal Cord Stimulation on Progressive Supranuclear Palsy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Our study hasn't been funded so far, but we will continue this study in the future.
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Jian Wang, Professor of neurology, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2019-506
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Progressive Supranuclear Palsy; Spinal Cord Stimulation
MeSH Terms: conditions — Supranuclear Palsy, Progressive | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- spinal cord stimulation (Experimental): the spinal cord stimulation was performed and operated
  Interventions: Procedure: Spinal Cord Stimulation

INTERVENTIONS:
Procedure: Spinal Cord Stimulation — Spinal cord stimulation is a treatment that implants a electrode in posterior epidural space of patient's spinal canal to send mild electric current to stimulate conducting bundle of the posterior column of the spinal cord and posterior horn sensory neurons.

SUMMARY:
The study is an open-label, prospective, single-arm, unicentral (Huashan Hospital Department of Neurology/ Neurosurgery) and exploratory clinical trial. Subjects will be enrolled from Parkinson's disease and Movement Disorder specialized outpatient department of Neurology in Huashan Hospital and network platform of chronic diseases. Spinal Cord Stimultion (SCS) will be performed in department of Neurosurgery and cerebral metabolism will be assessed in PET center of Huashan Hospital. Specialists in Neurology will follow up 3 months to record any unsafe incidents of progressive supranuclear palsy patients after the SCS surgery to evaluate safety. Meanwhile, improvement in gait disorder (including 10MWT and TUG test score) will be measured to evaluate efficacy.

DETAILED DESCRIPTION:
The Study to Evaluate the Safety and Efficacy of Spinal Cord Stimulation on Progressive Supranuclear Palsy is an open-label, prospective, single-arm, unicentral and exploratory clinical trial.

In the screening stage, patients clinically and radiologically diagnosed as progressive supranuclear palsy with prominent gait disturbance will be enrolled. Then comprehensive evaluations and spinal cord stimulation will be performed on patients eligible for stimulation. In the subsequent process of neuromodulation, changes of clinical presentations and cerebral metabolism of participants will be assessed. Any unsafe incidents in process will be recorded in detail.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis is Progressive Supranuclear Palsy according to International Movement Disorder society criteria for Progressive Supranuclear Palsy (2017).

2.18FDG-PET imaging was completed within three months before the operation, and the imaging results were consistent with characteristics of Progressive Supranuclear Palsy, supporting the clinical diagnosis of Progressive Supranuclear Palsy.

3. The clinical manifestation is prominent gait balance disorder with "freezing gait", "turn difficulties" and "feet like a stick on the ground", "instabillity" and a fall history in the nearly 6 months (fall number less than or equal to 3 times).Or the researchers observe the existence of gait balance disorder, but patients can still walk without using external things with new freezing gait questionnaire survey more than 1 minute.

4.Those who fully understand the research and sign the informed consent.

Exclusion Criteria:

1. Severe mental symptoms or depression state.
2. Severe cognitive dysfunction with MMSE less than 20.
3. Severe loss of postural reflexes (inability to stand and work independently) and depend on a walker or wheelchair.
4. Depend on nasal feeding tube.
5. Female in pregnant state when grouped.
6. Clear and definite history of neurological diseases (stroke, trauma, tumor, hydrocephalus.
7. Complicated with severe heart, liver or renal diseases.
8. Clear and definite contraindications for surgery, electrical stimulation and PET examination.
9. Unsuitable for surgery according to evaluation before the surgery.
10. Other conditions that researchers think unsuitable surgery.
11. Those who participant in other clinical trials at the same time.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Safety of Spinal Cord Stimulation | 3 months
  Safety evaluation will be performed 3 months after Spinal Cord Stimualtion
Efficacy of Spinal Cord Stimulation on walk gait. | 3 months after Spinal Cord Stimualtion.
  The change of 10 Meter Walk Test (10MWT) scores. The 10MWT recorded the time to finish the test, and the maximum time is 5 minutes. The longer time suggest more severe condition.
Efficacy of Spinal Cord Stimulation on walk time. | 3 months after Spinal Cord Stimualtion.
  Changes of the Time Up & Go (TUG) test score. TUG test recorded the time to finish the test, the minimum time is 0 and the maximum time is 5 minutes. The longer time suggest more severe condition.

SECONDARY OUTCOMES:
Alteration of cerebral metabolism in 18F-FDG-PET imaging | 6 months
  Alteration of cerebral metabolism in 18F-FDG-PET imaging 6 months after Spinal Cord Stimualtion
Alteration of gait, balance and motor score | 1 month, 6 months
  Alteration of gait, balance and motor score 1 month, 6 months after Spinal Cord Stimualtion. The New Freezing of Gait Questionnaire (NFOG-Q) will be assessed, with the minimum score to be 0 and the maximum score to be 30 scores, with higher scores suggest more severe condition.

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Tao Liu, MD, Study Director — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China